CLINICAL TRIAL: NCT03768141
Title: International Study on the Outcomes of Liver Surgery - LiverGroup.Org
Brief Title: International Liver Surgery Outcomes Study
Acronym: LiverGroup
Status: Completed | Type: Observational
Sponsor: Royal Free Hospital NHS Foundation Trust (Other)
Collaborators: Hospital Miguel Servet (Other)
Responsible Party: Principal Investigator, Dimitri Raptis, Senior Clinical Fellow, Royal Free Hospital NHS Foundation Trust
Other Study IDs: v.1.3.2011.11.30
Record Dates: First submitted 2018-12-03; First posted 2018-12-07 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Liver Diseases
Keywords: Liver; Surgery; Outcomes; Snapshot; Collaborative; International
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Liver surgery: Any type of liver surgery
  Interventions: Procedure: Liver surgery

INTERVENTIONS:
Procedure: Liver surgery — All indications (including benign and living donor resections), all co-morbidities, open, laparoscopic or robotic, single wedge resections to extended liver resections, single or two-stage hepatectomies, procedures with liver volume enhancement such as portal vein embolization (PVE), portal vein ligation (PVL), "Associating Liver Partition and Portal vein Ligation for Staged hepatectomy" (ALPPS), resections involving cold perfusion (ex-situ and ante-situ)

SUMMARY:
This study was to designed to measure the true worldwide practice of liver surgery and associated outcomes by recruiting multiple international centres, committing to consecutive patient registration per surgeon and undergo rigorous data validation. It is hoped that these data will provide a more appropriate guide to inform surgeons and patients to assess which level of complexity should be routinely offered for high tumour burden and anatomically difficult scenarios.

DETAILED DESCRIPTION:
Liver surgery was associated with at least 10% mortality in the 1970's. The safety of liver surgery has dramatically improved since with a mortality of now around 1-2%. Individual centres postulate that a perioperative mortality close to 0% should be the standard of major liver resection. Despite these claims, epidemiological studies showed a mortality rate of 6%. Outcomes in liver surgery are likely influenced by indications, complexity, centre and surgeon skills, equipment, centre and surgeon experience. The aim of LiverGroup.org is to develop an international data set on the outcomes of liver resections among a large number of international surgeons. The 'collaborative' model for 'snapshot' clinical audit is now well established and such research is a novel approach for assessing current practice in a short period of time. The primary objective of the study is to provide a verified record of the true perioperative morbidity and mortality of a representative set of liver surgeons worldwide in 2019. Secondary objectives include risk factors for mortality and morbidity using multivariable regression models. Any surgeon performing liver resections is eligible to participate in LiverGroup.org. All consecutive cases will be included and there are no minimum patient numbers per centre. Liver transplantation is excluded. There will be 3 months of prospective patient enrolment and 3 months follow up within the 12-month frame, January to December 2019. All liver resections, all indications, as well as all co-morbidities will be included. Liver transplantation, imaging-guided ablations and liver biopsies are excluded.

ELIGIBILITY:
Inclusion Criteria:

* All indications (including benign and living donor resections)
* All co-morbidities
* Open, laparoscopic or robotic
* Single wedge resections to extended liver resections
* Single or two-stage hepatectomies
* Procedures with liver volume enhancement such as PVE, PVL, ALPPS.
* Resections involving cold perfusion (ex-situ and ante-situ)
* There are no exclusion criteria as related to indication, age or comorbidities.

Exclusion Criteria:

* Liver transplantation
* Imaging-guided liver ablation techniques alone
* Liver biopsies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any adult patient undergoing liver surgery.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Mortality rate | From operation until 90 days postoperatively
  Death

SECONDARY OUTCOMES:
Complication rate | From operation until 90 days postoperatively
  Postoperative complications according the the Clavien-Dindo classification, the "liver Failure, Ascites, Bile leakage, Infection, Bleeding" (FABIB) liver specific classification, as well as the novel Comprehensive Complications Index® (CCI® ).
Liver failure rate | From operation until 90 days postoperative
  Posthepatectomy liver failure will be assessed according to the FABIB Classification, the "International Study Group of Liver Surgery" (ISGLS) criteria as well as the 50-50 criteria up to 90 days postoperatively.
Hospital stay | From operation until discharge from the hospital or up to 90 days postoperatively.
  The length of hospital stay is defined as the duration of hospitalization from the day of the operation until the day of discharge from the hospital.
Re-hospitalisation rate | From operation until 90 days postoperatively
  Readmission to any hospital

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Malagò, MD, PhD, Principal Investigator — Royal Free Hospital, London, UK
Locations (2):
- University of Zaragoza, Spain, Zaragoza, Spain
- Royal Free Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated and analysed during the current study will be available upon request from the Management Committee of LiverGroup.org. The study Primary Investigators will act as the custodians of the data. The data, however, belong to all collaborators. The Steering and Management committees together will decide after the publication of the main report about requests regarding secondary analysis and will consider all such requests based on quality and the validity of the proposed project and decide by majority decision. All data provided will be fully anonymized without any patient identifiers.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will become available after the completion and publication of the first study generated by LiverGroup.org
Access Criteria: The steering and management committees together will decide after the publication of the main report about requests regarding secondary analysis and will consider all such requests based on quality and the validity of the proposed project and decide by majority decision.
URL: https://livergroup.org/?q=protocol_full_version

REFERENCES:
- [Derived] LiverGroup.org Collaborative*. Outcomes of elective liver surgery worldwide: a global, prospective, multicenter, cross-sectional study. Int J Surg. 2023 Dec 1;109(12):3954-3966. doi: 10.1097/JS9.0000000000000711. PMID 38258997
- See also: Cloud Graphical User Interface for R Statistics - Statistical software for data analysis — http://www.rBiostatistics.com

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-30): https://cdn.clinicaltrials.gov/large-docs/41/NCT03768141/Prot_SAP_000.pdf